CLINICAL TRIAL: NCT00534859
Title: PROTECT I, A Prospective Feasibility Trial Investigating the Use of the IMPELLA RECOVER LP 2.5 System in Patients Undergoing High Risk PCI
Brief Title: PROTECT I, A Prospective Feasibility Trial Investigating the Use of IMPELLA RECOVER LP 2.5 System in Patients Undergoing High Risk PCI
Acronym: PROTECT I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Carol Pekar/Director of Clinical and Regulatory Affairs, Abiomed Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G050017
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Patients Undergoing High Risk PCI.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: High Risk PCI — High Risk Percutaneous Coronary Intervention

SUMMARY:
The objective of this feasibility study is to demonstrate that the device is safe and potentially efficacious for use in patients undergoing high risk Percutaneous Coronary Interventions(PCI).Patients will be enrolled if they meet inclusion & exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Non emergent PCI of at least one de novo or restenotic lesion in a native coronary vessel or bypass graft
* EF <35%

Exclusion Criteria:

* ST Myocardial Infarction
* Cardiac Arrest
* Cardiogenic Shock
* Thrombus Left Ventricle

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
MACCE Events at 30 days or discharge, whichever is longer | 30 days or discharge
  Major Adverse Cardiac and Cerebral (MACCE) events defined as death, new myocardial infarction, target vessel revascularization, urgent coronary artery bypass grafting procedure or cerebral vascular accident during and up to 30 days post-device explant or hospital discharge, whichever is longer.
Freedom from Hemodynamic compromise during PCI procedure | During procedure
  Freedom from Hemodynamic compromise during PCI procedure defined as: Mean Arterial Pressure (MAP) not falling below 60mm Hg for more than 10 minutes during the PCI procedure and additional pressor medication is not required

SECONDARY OUTCOMES:
Other intra-procedural and peri-procedural adverse events | During treatment and out to 90 days
Freedom from Ventricular fibrillation and Tachycardia requiring electrical cardioversion | During procedure
  Freedom from the following procedural-related events:
  i. Ventricular fibrillation ii. Tachycardia requiring electrical cardioversion
Angiographic Success | Post-PCI
  Angiographic success defined as residual stenosis <30% after stent implantation or <50% after balloon angioplasty.

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, M.D., Principal Investigator — Not affiliated with Abiomed
Locations (10):
- United States (9):
  - Scripps, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mass General Hospital, Boston, Massachusetts
  - Brigham & Womens, Boston, Massachusetts
  - William Beaumont, Royal Oak, Michigan
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Texas Heart, Houston, Texas
- Academic Medical Center, Amsterdam, Netherland, Netherlands

REFERENCES:
- [Derived] Dixon SR, Henriques JP, Mauri L, Sjauw K, Civitello A, Kar B, Loyalka P, Resnic FS, Teirstein P, Makkar R, Palacios IF, Collins M, Moses J, Benali K, O'Neill WW. A prospective feasibility trial investigating the use of the Impella 2.5 system in patients undergoing high-risk percutaneous coronary intervention (The PROTECT I Trial): initial U.S. experience. JACC Cardiovasc Interv. 2009 Feb;2(2):91-6. doi: 10.1016/j.jcin.2008.11.005. PMID 19463408